CLINICAL TRIAL: NCT02194257
Title: Investigation of the Metabolism and Pharmacokinetics of an Open Label Single Dose of 20 mg Ambroxol Administered as a Lozenge Together With an Oral Solution of 0.4 mg [14C]-Ambroxol in Healthy Male Volunteers
Brief Title: Investigation of the Metabolism and Pharmacokinetics of Ambroxol in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18.494
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- [14C]-cyclohexane ambroxol oral solution + ambroxol lozenge (Experimental)
  Interventions: Drug: [14C]-cyclohexane ambroxol oral solution; Drug: Ambroxol lozenge
- [14C]-benzyl ambroxol oral solution + ambroxol lozenge (Experimental)
  Interventions: Drug: [14C]-benzyl ambroxol oral solution; Drug: Ambroxol lozenge

INTERVENTIONS:
Drug: [14C]-cyclohexane ambroxol oral solution
  Arms: [14C]-cyclohexane ambroxol oral solution + ambroxol lozenge
Drug: [14C]-benzyl ambroxol oral solution
  Arms: [14C]-benzyl ambroxol oral solution + ambroxol lozenge
Drug: Ambroxol lozenge

SUMMARY:
Study to determine the basic pharmacokinetics of ambroxol and [14C]-radioactivity including mass balance, excretion pathways and complete metabolism in healthy male volunteers following administration of a lozenge of 20 mg ambroxol together with an oral solution of 0.4 mg [14C]-ambroxol labelled in two different positions

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and ≤65 years
* Body mass index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to study drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within ten days prior to administration until after the last sample from Visit 2 is collected
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during the stay in the trial centre
* Alcohol abuse (more than on average two units of alcoholic beverages per day or more than 14 units per week (one unit equals one pint [285 mL] of beer or lager, one glass [125 mL] of wine, 25 mL shot of 40% spirit)).
* Drug abuse
* Blood donation (more than 100 mL within 60 days prior to study drug administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the Trial until follow-up examination)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)

Exclusion criteria specific for this study:

* Veins unsuitable for blood sampling
* PR interval >220 ms or QRS interval >120 ms
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), during work or during participation in a medical trial in the previous year
* Irregular defecation pattern (less than once per two days)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Individual time course profiles of [14C]-radioactivity (in nmoleq/L or nmoleq/kg for faeces) in plasma | up to 120 hours after drug administration
Individual time course profiles of ambroxol in plasma | up to 120 hours after drug administration
Rate and extent of excretion mass balance based on the total radioactivity in urine and faeces | up to 216 hours after drug administration
Identification of major metabolites in urine, feces and plasma in comparison with various animal species | up to 48 hours after drug administration
Cblood cells/Cplasma ratio of [14C]-radioactivity and Cblood /Cplasma ratio of [14C]-radioactivity | up to 120 hours after drug administration
Cmax (maximum concentration of the analyte(s) in plasma) | up to 120 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte(s) in plasma) | up to 120 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 120 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte(s) in plasma over the time interval from 0 to infinity) | up to 120 hours after drug administration
λz (terminal rate constant in plasma) | up to 120 hours after drug administration
t1/2 (terminal half-life of the analyte(s) in plasma) | up to 120 hours after drug administration
MRTpo (mean residence time of the analyte(s) in the body after oral administration) | up to 120 hours after drug administration
CL/F (total clearance of the analyte in plasma after oral administration) | up to 120 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an oral dose) | up to 120 hours after drug administration
Ae0-tz (amount of analyte that is eliminated in urine within the time interval zero to tz) | up to 216 hours after drug administration
Aefaeces,0-tz (amount of analyte excreted in faeces within the time interval zero to tz) | up to 216 hours after drug administration
fefaeces,0-tz (fraction of analyte excreted in faeces within the time interval zero to tz in % of dose) | up to 216 hours after drug administration
CLR,t1-t2 (renal clearance of analyte from the within the time interval t1 to t2) | up to 216 hours after drug administration
fe0-tz (fraction of analyte excreted in urine within the time interval zero to tz in % of dose) | up to 216 hours after drug administration
Individual time course profiles of [14C]-radioactivity (in nmoleq/L or nmoleq/kg for faeces) in urine | up to 216 hours after drug administration
Individual time course profiles of [14C]-radioactivity (in nmoleq/L or nmoleq/kg for faeces) in faeces | up to 216 hours after drug administration
Individual time course profiles of ambroxol in urine | up to 216 hours after drug administration

SECONDARY OUTCOMES:
Number of patients with clinically significant changes vital signs (blood pressure [BP], pulse rate [PR]) | up to 39 days
Number of patients with adverse events | up to 39 days
Number of patients with clinically significant changes in 12-lead electrocardiogram (ECG) | up to 39 days
Number of patients with abnormal changes in laboratory parameters | up to 39 days
Assessment of tolerability on a 4-point scale | Day 14